CLINICAL TRIAL: NCT03282721
Title: Transverse Facial Cleft (Macrostomia) Repair: Modification of a Traditional Technique
Brief Title: Transverse Facial Cleft Repair Using Precise Location of Commissure
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Lian Zhou, Prof., Peking Union Medical College Hospital
Other Study IDs: S-K338
Record Dates: First submitted 2017-09-01; First posted 2017-09-14 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Transverse Facial Cleft

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- redesigned: the commissure constructions of the cleft side were precised located, include the upper and lower inherent vermilion border, the interior commissure, the outline of commissure, the exterior commissure, the upper skin-mucosa junction and the lower skin-mucosa junction.
  Interventions: Procedure: precise location of commissure
- classical: follows the simple-symmetry rule, the commissure of the healthy side is measured, and then the affected side is located accordingly.

INTERVENTIONS:
Procedure: precise location of commissure
  Groups: redesigned

SUMMARY:
To compare the effect of redesigned transverse facial cleft treatment and traditional transverse facial cleft treatment.

DETAILED DESCRIPTION:
Nine patients with transverse facial cleft were treated with redesigned repair using precise location of commissure. The main outcome measurement included scar, symmetry of the commissure. They were graded in five scores by five resident physicians who had never seen the patients. The results were compared with healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of transverse facial cleft disease;
* Must not received any lip surgeries before;
* Such disease can be accompanied by external ear abnormalities, hypoplastic mandible, cleft lip and palate.

Exclusion Criteria:

* Severe general diseases;
* Patients who had been treated with lip surgery;
* Patients and/or his/her family didn't want to continue the clinical trial.

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients diagnosed with transverse facial cleft who hadn't receive any treatment.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2016-01-30 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Scar of the repaired commissures | 6 to 12 months after surgery
  scar of the repaired commissures was graded in five points. They were scored by five resident physicians who had never seen the patients.
symmetry of the commissures | 6 to 12 months after surgery
  symmetry of the commissures was graded in five points. They were scored by five resident physicians who had never seen the patients.

SECONDARY OUTCOMES:
scar of the repaired commissures | immediately after surgery
  scar of the repaired commissures was graded in five points. They were scored by five resident physicians who had never seen the patients.
symmetry of the commissures | immediately after surgery
  symmetry of the commissures was graded in five points. They were scored by five resident physicians who had never seen the patients.
scar of the repaired commissures | 1 to 6 months after surgery
  scar of the repaired commissure was graded in five points. They were scored by five resident physicians who had never seen the patients.
symmetry of the commissures | 1 to 6 months after surgery
  symmetry of the commissures was graded in five points. They were scored by five resident physicians who had never seen the patients.

CONTACTS AND LOCATIONS:
Overall Officials: LIAN ZHOU, D.D.S, Principal Investigator — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: No